CLINICAL TRIAL: NCT05197543
Title: Biomechanical Rupture Risk Assessment in Management of Patients With Abdominal Aortic Aneurysm in COVID-19 Pandemic
Brief Title: AAA Rupture Risk Assessment in COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Masaryk University (Other)
Collaborators: VSB - Technical University of Ostrava (Unknown)
Responsible Party: Principal Investigator, Luboš Kubíček, Principal Invastigator, Masaryk University
Other Study IDs: BRRA19
Record Dates: First submitted 2022-01-15; First posted 2022-01-19 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Abdominal Aortic Aneurysm; COVID-19
Keywords: Abdominal aortic Aneurysm; Biomechanics; Rupture risk; Predictability; COVID-19
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BRRA group: Rupture risk of asymptomatic AAAs in this group was estimated using Biomechanical rupture rist assessment (BRRA). BRRA considers an AAA as a pressure vessel and estimates its risk of rupture by comparing its wall stress to wall strength
  Interventions: Diagnostic Test: Biomechanical rupture risk assessment
- Maximal diameter group: Rupture risk of asymptomatic AAAs in this group was estimated by a classical approach based on a maximal diameter.

INTERVENTIONS:
Diagnostic Test: Biomechanical rupture risk assessment — 3D computational model is created from CT angiographic images available during standard AAA diagnostic process. Vascular wall stress is assessed based on the 3D model using Finite element method to identify highly stressed parts of AAA and results are compared to populational wall strength information (gathered from previous large histological study), thus rupture risk (stress/strength ratio) of each particular AAA is estimated. Other relevant factors such as gender, blood pressure, presence of intraluminal thrombus etc. are used during the calculation as well.
  Other Names: Vascular wall stress assessment using finite element method
  Groups: BRRA group

SUMMARY:
The acute phase of the COVID-19 pandemic requires a redefinition of healthcare system to increase the number of available intensive care units for COVID-19 patients. This leads to the postponing of elective surgeries including the treatment of abdominal aortic aneurysm (AAA). The probabilistic rupture risk index (PRRI) recently showed its advantage over the diameter criterion in AAA rupture risk assessment. Its major improvement is in increased specificity and yet has the same sensitivity as the maximal diameter criterion. The objective of this study was to test the clinical applicability of the PRRI diagnostic method in a quasi-prospective observational patient cohort study.

ELIGIBILITY:
Inclusion Criteria:

* presence of asymptomatic abdominal aortic aneurysm (AAA)
* regular CT angiography scans available

Exclusion Criteria:

* rupture of AAA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with asymptomatic AAA during the COVID-19 pandemic period. During this period an elective surgeries had to be posponed and there was a need for auxiliary diagnostic method able to identify AAAs with high risk of rupture.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Test the clinical applicability of the BRRA method | 21 months
  Identify the number of number of false positive and false negative cases assessed by BRRA method according to clinical data and compare these data to control group where the decision making process was based only on maximal diameter of AAA

SECONDARY OUTCOMES:
Reduction of time required for AAA assessment | 21 months
  To investigate the feasibility of cooperation between the biomechanical and medical teams in a modified AAA management workflow leading to reduced time required for an AAA assessment

CONTACTS AND LOCATIONS:
Overall Officials: Robert Staffa, M.D., Ph.D., Study Director — Masaryk University
Locations (1):
- St. Anne´s University Hospital in Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
All data are stored in standard patient documentation in study center, anonymized data can be shared on request